CLINICAL TRIAL: NCT04572750
Title: Promoting Benzodiazepine Cessation Through an Electronically-delivered Patient Self-management Intervention
Acronym: EMPOWER-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 18-026
Record Dates: First submitted 2020-08-20; First posted 2020-10-01 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Taking Benzodiazepines for Any Reason for 3 Months; Benzodiazepine Dependence
Keywords: insomnia; anxiety; benzodiazepine; self-help; patient education; electronic intervention
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The EMPOWER-ED intervention is an app that runs on a smart phone or computer. It will provide education about the risk of benzodiazepine, a tool to create a method of self-tapering, and information on how to succeed at reducing or quitting benzodiazepine use. Individuals in the treatment condition of the trial will be given access to EMPOWER-ED on any platform they wish to use.
Who Masked: Outcomes Assessor
Masking Description: At follow-up interview, the interviewer will no know whether the individual was in the treatment or control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EMPOWER-ED (Experimental): Individuals will be given access on their preferred platform to an electronic self-help app focused on reducing benzodiazepine use
  Interventions: Behavioral: EMPOWER-ED
- Control (No Intervention): Individuals will be provided care as usual

INTERVENTIONS:
Behavioral: EMPOWER-ED — An electronic app that runs on a variety of platforms and provides education and tools designed to promote self-driven reduction of benzodiazepines.
  Arms: EMPOWER-ED

SUMMARY:
Benzodiazepines (e.g., Ativan, Xanax) are widely prescribed medications that are used mainly to treat anxiety and sleeping difficulties. Long-term use of benzodiazepine carries risks of physical dependence, addiction, falls and other accidents, and problems in thinking/concentrating. Researchers in Canada developed a printed self-help packet that enabled many individuals to reduce or cease taking benzodiazepines on their own. This study is designed to tailor that packet to the Veteran population, convert it to an app that people can use on their laptop or smart phone, and test whether the app helps promote benzodiazepine prescribing.

DETAILED DESCRIPTION:
Background: Long-term use of benzodiazepine medication has been increasing sharply inside and outside of VA, raising the risk of cognitive decline, falls, and overdose among patients. A self-directed benzodiazepine tapering intervention known as EMPOWER was shown effective in a non-VA clinical trial, and within VA there is significant interest in tailoring it to and providing it for Veterans. Significance: Although often useful as short-term medications, when taken for extended periods benzodiazepines carry risk of cognitive decline and other brain damage, falls and other accidents, benzodiazepine dependence and opioid-benzodiazepine overdose (VA Pharmacy Benefits Management Academic Detailing Service, 2017). This is major concern within VA, which prescribes benzodiazepines to over 350,000 Veterans a year, 2/3 of whom take them long-term (i.e., 3 months or more) (VA Pharmacy Benefits Management Academic Detailing Service, 2017). Innovation: Because the EMPOWER intervention was paper-and-pencil based, it would be useful to convert it to an electronic version that worked on smart phones, tablets, and/or desktop computers. Accordingly, the proposed project intends to convert EMPOWER to electronic format and to tailor it to the needs and preferences of the Veteran population. Specific Aims: Aim 1: Tailor a promising non-VA benzodiazepine cessation intervention (EMPOWER) to Veterans and simultaneously convert it from paper-and-pencil to electronic format. Aim 2: Conduct a randomized clinical trial of the effectiveness of the tailored, electronic intervention (EMPOWER-ED) on VA primary care patients' benzodiazepine cessation/reduction and functional outcomes. Aim 3: Conduct a budget impact analysis to estimate the costs of implementing the EMPOWER-ED throughout VA. Methodology: This conversion and tailoring will be an iterative process that the project team will conduct via focus groups comprising Veterans, VA primary care providers, and VA operational partners. When the revised intervention, called EMPOWER-ED (for EMPOWER "Electronically Delivered"), is fully designed and has been successfully beta-tested by Veterans, its effectiveness will be evaluated in a randomized clinical trial with 170 Veterans who have been on benzodiazepines for at least 3 months. The primary hypothesis of the study is that those receiving EMPOWER-ED will be significantly more likely than controls to cease benzodiazepines entirely, and, to reduce their dose by at least 25%, at 6-month follow-up. The secondary hypothesis is that Veterans receiving EMPOWER-ED will also experience fewer anxiety symptoms, better sleep quality, and overall health/quality of life at 6-month follow-up. A supplemental analysis of benzodiazepine use only will be conducted using VA databases at 12 months to evaluate whether changes identified at 6 months persist over time. The VA operational partners of the project team (Pharmacy Benefits Management, Psychotropic Drug Safety Initiative, and Office of Connected Care) are committed to disseminating EMPOWER-ED if it proves successful. Therefore, a third aim of the study is to undertake a budget impact analysis to determine what the costs would be to implement EMPOWER-ED in the VA systemwide. Next Steps/Implementation: Because electronically-delivered interventions are inexpensive to disseminate once they have been developed, this project has an excellent chance to promote health care value by creating an easily scaled-up, method of reducing the prevalence of a widespread risk to Veterans' health.

ELIGIBILITY:
Inclusion Criteria:

* Veterans having a VA primary care provider and taking prescribed benzodiazepines for at least 3 months
* Have access to a smartphone, tablet, or computer

Exclusion Criteria:

* Individuals diagnosed with schizophrenia, dementia, seizure disorder, and/or spinal cord injury
* Individuals receiving palliative care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith N. Humphreys, PhD MA, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA; Michael A Cucciare, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System , Little Rock, AR
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cucciare MA, Abraham TH, Kemp L, White P, Marchant K, Hagedorn HJ, Humphreys K. Adapting the Eliminating Medications Through Patient Ownership of End Results Protocol to Promote Benzodiazepine Cessation Among US Military Veterans: Focus Group Study With US Military Veterans and National Veterans Health Administration Leaders. J Med Internet Res. 2022 Sep 19;24(9):e35514. doi: 10.2196/35514. PMID 36121697
- [Result] Cucciare MA, Hagedorn HJ, Bounthavong M, Abraham TH, Greene CJ, Han X, Kemp L, Marchant K, White P, Humphreys K. Promoting benzodiazepine cessation through an electronically-delivered patient self-management intervention (EMPOWER-ED): Randomized controlled trial protocol. Contemp Clin Trials Commun. 2022 Sep 5;29:100994. doi: 10.1016/j.conctc.2022.100994. eCollection 2022 Oct. PMID 36111174
- [Derived] Humphreys K, Hagedorn H, Han X, Kemp L, Poitra N, Cucciare MA. Electronic Intervention for Patient-Managed Benzodiazepine Tapering: A Randomized Clinical Trial. JAMA Netw Open. 2026 Jan 2;9(1):e2551807. doi: 10.1001/jamanetworkopen.2025.51807. PMID 41533380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 484 individuals were approach about the study, and 170 participants were enrolled. 244 individuals were not interested and 70 were ineligible.
Period: Overall Study
Arm/Group | EMPOWER-ED | Control
Started | 85 | 85
Completed | 82 | 79
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Population: Data not available for 9 participants due to ineligibility
Groups:
- Total: Total of all reporting groups
Arm/Group | EMPOWER-ED | Control | Total
Number analyzed (Participants) | 82 | 79 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] — The minimum and the maximum are 27 and 94 respectively.
  years | 62.28 (13.58) | 61.48 (13.88) | 61.89 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 16 | 27
  Male | 71 | 63 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 6 | 11
  White | 75 | 68 | 143
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: 25% Reduction in Benzodiazepine Use
Description: This outcome reflects an individual cutting their dose of benzodiazepine medication by one quarter or more
Time Frame: 6 months
Population: We excluded nine patients because they were not eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | EMPOWER-ED | Control
Number analyzed (Participants) | 82 | 79
Participants | 14 | 6

2. Primary Outcome: Cessation of Benzodiazepine Use
Description: This outcome reflects an individual eliminating their benzodiazepine use from baseline to 6 month follow-up
Time Frame: 6 Months
Population: We excluded nine subjects because they were not eligible.
Measure: Count of Participants; unit: Participants
Arm/Group | EMPOWER-ED | Control
Number analyzed (Participants) | 82 | 79
Participants | 10 | 2

3. Secondary Outcome: Anxiety
Description: Anxiety at baseline and 6-month follow-up will be measured using Spitzer's 7 item generalized anxiety disorder subscale. The minimum and the maximum of the measure are 0 and 21 respectively with higher score representing anxiety symptoms occurred more frequently.
Time Frame: Baseline, 6 months
Population: We excluded nine subjects because they were not eligible.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EMPOWER-ED | Control
Number analyzed (Participants) | 82 | 79
units on a scale
  baseline | 9.77 (9.17) | 8.86 (8.81)
  follow-up | 8.23 (6.60) | 7.26 (6.33)

4. Secondary Outcome: Sleep Quality
Description: This outcome measures sleep quality as assessed by the Patient-Reporter Outcomes Measurement System. The minimum and the maximum of the measure are 8 and 40 respectively with higher score representing worse quality of sleep.
Time Frame: Baseline, 6 months
Population: We excluded nine patients because they were not eligible.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EMPOWER-ED | Control
Number analyzed (Participants) | 82 | 79
units on a scale
  baseline | 23.84 (12.02) | 24.53 (13.87)
  6-month follow-up | 23.80 (8.54) | 23.64 (7.86)

5. Secondary Outcome: Overall Health and Quality of Life
Description: Overall health and quality of life (Physical Component Summary and Mental Component Summary) will be assessed using the RAND Veterans SF-12. The minimum and the maximum of the physical component summary measure are 8.66 and 64.91 respectively with higher score representing better physical functioning. The minimum and the maximum of the mental component summary measure are 14.91 and 70.61 respectively with higher score representing better mental functioning.
Time Frame: Baseline, 6 months
Population: We excluded nine patients because they were not eligible.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EMPOWER-ED | Control
Number analyzed (Participants) | 82 | 79
units on a scale
  Baseline Physical Component Summary | 38.06 (15.84) | 38.03 (19.07)
  Follow-up Physical Component Summary | 37.45 (10.77) | 37.26 (13.03)
  Baseline Mental Component Summary | 40.19 (18.99) | 40.21 (17.25)
  Follow-up Mental Component Summary | 40.65 (11.64) | 41.27 (10.24)

ADVERSE EVENTS:
Time Frame: from enrollment until 6-month follow-up
Arm/Group | EMPOWER-ED | Control
All-Cause Mortality (participants affected / at risk) | 0/85 | 2/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 0/85 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04572750/Prot_SAP_001.pdf
  • Informed Consent Form (2022-09-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04572750/ICF_000.pdf